CLINICAL TRIAL: NCT02535663
Title: Consumption of Dairy Yogurt With Rhamnogalacturonan in Korean Citrus Hallabong Peel Polysaccharide Enhanced Immune Function and Attenuated Inflammatory Response
Brief Title: Consumption of Dairy Yogurt Enhanced Immune Function
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: YF_immune
Record Dates: First submitted 2015-08-26; First posted 2015-08-28 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Healthy Volunteers
Keywords: rhamnogalacturonan; Natural killer cell activity; interleukin-12; interferon-gamma; immune function; inflammatory

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- test group (Experimental): Dietary Supplement: RG consumed one pack (150ml) of dairy yogurt containing RG (100mg Korean citrus Hallabong peel polysaccharide) per day for 8 weeks
  Interventions: Dietary Supplement: RG
- placebo (Placebo Comparator): Dietary Supplement: placebo consumed one pack (150ml) of dairy yogurt without RG per day for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: RG — The 100mg Korean citrus Hallabong peel polysaccharide contained 60mg rhamnogalacturonan (RG), 20mg mono- and di-saccharide, 5mg polyphenol, 5mg ash and 10mg moisture
  Arms: test group
Dietary Supplement: Placebo — Same product without RG
  Arms: placebo

SUMMARY:
To investigate the impact of consumption of dairy yogurt with rhamnogalacturonan (RG) in Korean citrus Hallabong peel polysaccharide on Natural Killer (NK) cell activity and circulating cytokine levels.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study was conducted on 120 nondiabetic and nonobese subjects. Over an 8 week period, the test group consumed one pack (150ml) of dairy yogurt with 50mg probiotics and 100mg Korean citrus Hallabong peel polysaccharide (60% RG, 20% mono- and di-saccharide, 5% polyphenol) each day, whereas the placebo group consumed the same product without Korean citrus Hallabong peel polysaccharide. NK cell activities (%) were measured based on the ratios of effector cells (E) (peripheral blood mononuclear cell, PBMC) from each participant to Target cell (T) (K562 cells) as 10:1, 5:1, 2.5:1 or 1.25:1.

ELIGIBILITY:
Inclusion Criteria:

* The levels of white blood cells under 8x10^3/μL
* males and females
* 30-69 years old
* nondiabetic and nonobese subjects
* able to give informed consent

Exclusion Criteria:

* consumption of any probiotic products within 1 month before screening
* unstable body weight (body-weight change > 2 kg within 3 months before screening)
* diabetes
* history/presence of significant metabolic disease
* pregnancy or breast-feeding
* acute or chronic infection
* liver disease, kidney disease, gastrointestinal disease, or any other acute or chronic disease requiring treatment
* subjects taking any drugs or supplements

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
serum cytokine concentrations | change from baseline in RG at 8 weeks
  Primary outcome will be tested before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Ho Lee, PhD, Principal Investigator — Yonsei University
Locations (1):
- Yonsei University, Seoul, South Korea

REFERENCES:
- [Derived] Lee MH, Kim M, Kim M, Kwak JH, Chang DH, Yu WK, Lee SH, Lee JH. Consumption of dairy yogurt with the polysaccharide rhamnogalacturonan from the peel of the Korean citrus hallabong enhances immune function and attenuates the inflammatory response. Food Funct. 2016 Jun 15;7(6):2833-9. doi: 10.1039/c5fo01103e. PMID 27225729